CLINICAL TRIAL: NCT06836102
Title: The Potential of Nano-based Gel of Orange Peel Extract in Management of Epistaxis : a Randomized Double Blind Clinical Study
Brief Title: Usage of Orange Peel Extract in Management of Epistaxis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mostafa Nasr Zayed, lecturer of otorhinolaryngology Minia university, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: orange peel in epistaxis
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- gel of Orange peel extract (Active Comparator): usage of gel of Orange peel extract as a local treatment of epistaxis
  Interventions: Dietary Supplement: Orange
- nano-based gel of Orange peel extract (Active Comparator): usage of nano-based gel of Orange peel extract as a local treatment of epistaxis
  Interventions: Dietary Supplement: Orange
- placebo (Placebo Comparator): usage of placebo in control cases
  Interventions: Dietary Supplement: Orange

INTERVENTIONS:
Dietary Supplement: Orange — usage of orange peel extract in gel layer in treatment of epistaxis

SUMMARY:
Efficacy of orange peel extract in treatment of epistaxis in children

DETAILED DESCRIPTION:
Formulation of orange peel extract into gel substance and usage of it in local treatment of epistaxis

ELIGIBILITY:
Inclusion Criteria:

* children with anterior epistaxis from little's area

Exclusion Criteria:

* patient with nasal polyp.
* patients with hematological abnormalities.
* patients with general diseases affecting coagulation system.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The potential of nano-based gel of Orange peel extract in management of epistaxis | From enrollment to the end of treatment at 4 weeks
  assessment of epistaxis ( amount, severity and frequency ) according to ESS ( Epistaxis Severity Score ) between patients in study groups

IPD SHARING:
Plan to Share IPD: Yes
result
Supporting Information: ICF, CSR
Time Frame: 3 months
Access Criteria: contact by emailing
URL: http://drmostafanasr1988@gmail.com

REFERENCES:
- [Background] Andrade MA, Barbosa CH, Shah MA, Ahmad N, Vilarinho F, Khwaldia K, Silva AS, Ramos F. Citrus By-Products: Valuable Source of Bioactive Compounds for Food Applications. Antioxidants (Basel). 2022 Dec 25;12(1):38. doi: 10.3390/antiox12010038. PMID 36670900
- See also: Epistaxis: Outpatient Management — https://www.aafp.org/pubs/afp/issues/2018/0815/p240.html
- Available data/document: Study Protocol: drmostafanasr1988@gmail.com — https://doi.org/10.1016/j.hermed.2021.100468